CLINICAL TRIAL: NCT00245648
Title: Female Sex is an Independent Predictor of Death and Bleeding Among Fibrinolytic Treated Patients With AMI; Results of the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries - V Trial
Brief Title: Female Sex is an Independent Predictor of Death and Bleeding Among Fibrinolytic Treated Patients With AMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: The Cleveland Clinic (Other); Centocor, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Harmony R. Reynolds, Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GUSTOVsex
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Thrombolytic Therapy

INTERVENTIONS:
Drug: fibrinolytic therapy or combination reduced fibrinolytic therapy

SUMMARY:
This study evaluated differences between men and women in the presentation, management and outcome of heart attacks within the GUSTO V study.

DETAILED DESCRIPTION:
The Global Use of Strategies to Open Occluded Arteries in Acute Coronary Syndromes (GUSTO) V trial examined a large, contemporary cohort of women and men with ST elevation myocardial infarction (STEMI) treated with fibrinolytic therapy. The objective of the present study was to evaluate sex differences in presentation, management and outcome in GUSTO V.

ELIGIBILITY:
Inclusion Criteria:

* inclusion into GUSTO V

Exclusion Criteria:

* lack of availability of data (database study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 30 days
  All cause mortality at 30 days after randomization.

SECONDARY OUTCOMES:
Secondary Outcomes | 7 days
  Incidence of myocardial reinfarction as evidenced by new electrocardiographic changes or elevation in cardiac enzyme levels with recurrent chest pain within 7 days, bleeding, stoke, intracranial hemorrhage (ICH), and complications of MI.

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Topol EJ; GUSTO V Investigators. Reperfusion therapy for acute myocardial infarction with fibrinolytic therapy or combination reduced fibrinolytic therapy and platelet glycoprotein IIb/IIIa inhibition: the GUSTO V randomised trial. Lancet. 2001 Jun 16;357(9272):1905-14. doi: 10.1016/s0140-6736(00)05059-5. PMID 11425410
- [Background] Lincoff AM, Califf RM, Van de Werf F, Willerson JT, White HD, Armstrong PW, Guetta V, Gibler WB, Hochman JS, Bode C, Vahanian A, Steg PG, Ardissino D, Savonitto S, Bar F, Sadowski Z, Betriu A, Booth JE, Wolski K, Waller M, Topol EJ; Global Use of Strategies To Open Coronary Arteries Investigators (GUSTO). Mortality at 1 year with combination platelet glycoprotein IIb/IIIa inhibition and reduced-dose fibrinolytic therapy vs conventional fibrinolytic therapy for acute myocardial infarction: GUSTO V randomized trial. JAMA. 2002 Nov 6;288(17):2130-5. doi: 10.1001/jama.288.17.2130. PMID 12413372
- [Derived] Reynolds HR, Farkouh ME, Lincoff AM, Hsu A, Swahn E, Sadowski ZP, White JA, Topol EJ, Hochman JS; GUSTO V Investigators. Impact of female sex on death and bleeding after fibrinolytic treatment of myocardial infarction in GUSTO V. Arch Intern Med. 2007 Oct 22;167(19):2054-60. doi: 10.1001/archinte.167.19.2054. PMID 17954798